CLINICAL TRIAL: NCT04325750
Title: Effects of Capacitive and Resistive Energy Transfer Therapy in Pre and Post-treatment Medial Gastrocnemius in National Level Basketball Players
Brief Title: Energy Transfer Therapy in Treatment of Medial Gastrocnemius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Principal Investigator, Carlos Barrios Pitarque, PhD. Dean of Faculty of Medicine and Health Sciences, Fundación Universidad Católica de Valencia San Vicente Mártir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCV2017-2018-40
Record Dates: First submitted 2020-03-23; First posted 2020-03-30 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Strain of Gastrocnemius Muscle (Diagnosis); Diathermy Plate Burn; Thermography; Sports Physical Therapy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The simulated mode technique is applied (machine off)
  Interventions: Other: Placebo
- TECAR THERAPY (Experimental): The intervention will be performed with the T-Care TECAR® therapy machine at the latent trigger points of both gastrocnemius. The professional will apply the therapy with the generator that emits radio frequency signals of 0.5 MHz at a variable power with a maximum of 300W. The frequency to be used will be 500MHz with an intensity of 40% and with direct current.
  Interventions: Procedure: TECAR Therapy

INTERVENTIONS:
Procedure: TECAR Therapy — The intervention will be performed with the T-Care TECAR® therapy machine at the latent trigger points of both gastrocnemius. The professional will apply the therapy with the generator that emits radio frequency signals of 0.5 MHz at a variable power with a maximum of 300W. The frequency to be used will be 500MHz with an intensity of 40% and with direct current.
  Arms: TECAR THERAPY
Other: Placebo — simulated TECAR Therapy (machine off)
  Arms: Control

SUMMARY:
This study develops the effects of Capacitive and Resistive Energy Transfer Therapy (TECAR) on medial gastrocnemius using thermographic cameras, algometry and lunge tests, in a pre-post study with basketball players using a control group to which placebo is applied. (simulated technique) and an intervention group to which the technique is performed. The main objective of the study is to establish whether the TECAR produces physiological and mechanical changes in the subjects that improve muscle recovery.

ELIGIBILITY:
Inclusion Criteria:

* Male players
* Semi-professional players who are currently active
* Not have suffered a lower limb injury in the last 6 months before the study
* Not having suffered a rupture of the triceps surae
* Contain a latent trigger point in the medial gastrocnemius

Exclusion Criteria:

* Players suffering from any disease that could alter the study or be contradictory

Ages: 16 Years to 39 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 30 minutes
  Visual analogue scale (VAS) of pain

SECONDARY OUTCOMES:
Back flexion | 30 minutes
  LUNGE Test
Thermographic evaluation | 30 minutes
  Ymiko Wifi Digital Weather Station with FLIR E60 camera and interpreted with FLIR tools software.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Barrios, PhD, Study Director — Universidad Católica de Valencia San Vicente Mártir
Locations (1):
- Universidad Católica de Valencia San Vicente Mártir, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No